CLINICAL TRIAL: NCT02654587
Title: A Randomized Phase III Trial of OSE2101 Compared With Chemotherapy (Docetaxel or Pemetrexed) in HLA-A2 Positive Patients With Advanced Non-Small Cell Lung Cancer With Progressive Disease After Immune Checkpoint Inhibitors
Brief Title: OSE2101 Versus Chemotherapy in HLA-A2 Positive Patients With Advanced NSCLC After Immune Checkpoint Inhibitor Failure
Acronym: ATALANTE-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to COVID-19
Sponsor: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSE2101C301; 2015-003183-36 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced Non-Small-Cell Lung Cancer; Therapeutic Cancer Vaccine; Resistance to Immunotherapy; Quality of Life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — IDM 2101; Docetaxel; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Two-step open-label study with a planned interim OS futility in experimental arm per Fleming design (Step1) Central randomisation (2:1) with stratification by histology (non-squamous versus squamous), best response to first-line treatment [complete response (CR) or partial response (PR) versus stable disease (SD) or PD] and line of prior anti-PD(L)1 treatment (first-line when combined with platinum-based chemotherapy versus second-line when administered as sequential treatment after first-line platinum-based chemotherapy).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSE2101 (Experimental): OSE2101 was administered as a 1 mL-subcutaneous injection on Day 1 every three weeks for six cycles, then every eight weeks for the remainder of year one and finally every twelve weeks beyond year one until unequivocal RECIST 1.1-defined disease progression as determined by the investigator, unacceptable toxicity, or consent withdrawal. Should pseudo progression or delayed response to treatment suspected in arm A, investigator may continue treatment beyond the time of RECIST-defined progression, if the patient is perceived to be experiencing clinical benefit of OSE2101. OSE2101 dose was 5 mg of peptides (0.5 mg for each peptide).
  Interventions: Biological: OSE2101
- Docetaxel or Pemetrexed (Active Comparator): Patients receiving docetaxel: Docetaxel 75 mg/m2 will be administered by intravenous infusion over 1 hour on Day 1 of a 21-day cycle.
  Patients receiving pemetrexed: Pemetrexed, 500 mg/m2, will be administered by intravenous infusion over 10 minutes on Day 1 of a 21-day cycle.
  Docetaxel and pemetrexed will be continued until unequivocal RECIST 1.1-defined disease progression as determined by the investigator, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Biological: OSE2101
  Other Names: TEDOPI; EP-2101; EP2101; IDM-2101
  Arms: OSE2101
Drug: Docetaxel
  Other Names: Taxotere
  Arms: Docetaxel or Pemetrexed
Drug: Pemetrexed
  Other Names: Alimta
  Arms: Docetaxel or Pemetrexed

SUMMARY:
The aim of this clinical trial was to determine if the therapeutic cancer vaccine OSE2101 (TEDOPI) was more effective than standard chemotherapy (docetaxel or pemetrexed) in treating HLA-A2 positive patients with metastatic NSCLC who progressed after sequential or concurrent chemotherapy and immune checkpoint inhibitor given in first or second-line treatment.

The main questions were to compare the survival, the tolerance to treatment and the quality of life of patients between the two arms of treatment (OSE2101 versus standard chemotherapy)

DETAILED DESCRIPTION:
The study was a two-step randomized (2:1) study. Patients were stratified by histology (non-squamous versus squamous), best response to first-line treatment [complete response or partial response versus stable disease or progressive disease] and line of treatment with prior ICI (first-line ICI when combined with platinum-based chemotherapy versus second-line ICI when administered as sequential treatment). Primary endpoint was overall survival (OS). Interim OS futility analysis was planned as per Fleming design. In April 2020 at the time of the interim analysis, a decision was taken to early stop the accrual due to COVID-19 after 219 out of 363 patients were randomized. It led to a decrease of the study power from 80% to 62%. At the time of the interim analysis, a subgroup of patients was identified from stratification factor based on a clinical and biological rationale: those who received ICI second line and having received at least 12 weeks ICI. This subgroup was defined as ICI secondary resistance. The final analysis was carried out in the subgroup of patients with ICI secondary resistance and in all patients (ICI primary and secondary resistance).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Willingness and ability to comply with the clinical study procedures.
3. Female or male, 18 years of age or older
4. Histologically or cytologically proven diagnosis of Non-Small Cell Lung Cancer (NSCLC) that is locally advanced (stage III) unsuitable for radiotherapy or metastatic (stage IV) according to the 8th edition of tumor, node, metastasis (TNM) in Lung Cancer
5. Subjects with disease recurrence or progression after immune checkpoint inhibitor and platinum-based chemotherapy:

   i) either 1st line chemotherapy followed by 2nd line immune checkpoint inhibitor, or ii) 1st line combination of immune checkpoint inhibitor and chemotherapy Patients with progression during or within 12 months after the end of immune checkpoint inhibitor given as sequential or concomitant platinum-based chemotherapy ± radiation for locally advanced disease (stage III) were eligible
6. Subjects with measurable or non-measurable lesions according to RECIST 1.1
7. Subjects must express HLA-A2 phenotype (central test in blood)
8. Subjects must be considered suitable for chemotherapy with single-agent pemetrexed or single-agent docetaxel
9. Subjects with brain metastases were eligible if treated (whole brain radiotherapy, stereotaxic radiotherapy, surgery) at least 3 weeks prior to initiation of study treatment and have no symptoms related to brain metastases for at least 2 weeks before initiation of study treatment and are not taking any forbidden medications
10. Any prior chemotherapy, immunotherapy, hormonal therapy, radiation therapy or surgeries must have been completed at least 3 weeks prior to initiation of study treatment.
11. Any toxicity from prior therapy must have recovered to ≤ Grade 1 (except alopecia)
12. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
13. Adequate organ function as defined by all the following criteria:

    * Albuminemia > 25g/L
    * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 1.5 x upper limit of normal (ULN) with alkaline phosphatase ≤ 2.5 x ULN, or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to liver metastases
    * Total serum bilirubin ≤ 1.5 x ULN
    * Absolute neutrophil count (ANC) ≥ 1500/L
    * Platelets ≥ 100000/L
    * Hemoglobin ≥ 9.0 g/dL (in the absence of transfusion within 2 weeks before randomization)
    * Creatinine clearance (based on modified Cockcroft-Gault formula) ≥ 45 ml/min.

Exclusion Criteria:

1. Small-cell lung cancer/mixed NSCLC with small cell component or other neuroendocrine lung cancers (typical and atypical carcinoids, large-cell neuroendocrine carcinomas)
2. Patients with squamous cell carcinoma histology, and who had docetaxel as part of his prior chemotherapy
3. Current or previous treatment with investigational therapy in another therapeutic clinical trial (interrupted less than 4 weeks before study treatment initiation)
4. Patients whose tumor harbors EGFR gene mutation that sensitizes tumors to Tyrosine-Kinase Inhibitor (TKI) (EGFR exon 18-21) or Anaplastic Lymphoma Kinase (ALK) rearrangement
5. Ongoing immunotherapy (checkpoint inhibition, antigen immunotherapy that would be scheduled to continue concomitantly to the study)
6. Spinal cord compression (unless treated with the patient attaining good pain control and stable or recovered neurologic function), carcinomatous meningitis, or leptomeningeal disease
7. Patients with squamous cell histology or non-squamous cell histology previously treated by pemetrexed with a contraindication for docetaxel with grade ≥ 2 neuropathy or hypersensitivity reaction to medications formulated with polysorbate 80 (Tween 80)
8. Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
9. Treatment with corticosteroids in the last 3-week period before inclusion, except for topical, ocular, intra-articular, intranasal, and inhaled corticosteroids with minimal systemic absorption (e.g. with a dose ≤ 500 microgram beclomethasone equivalent for inhaled steroids), or steroid doses ≤ 10 mg daily prednisone equivalent which are permitted
10. A recognized immunodeficiency disease including human immunodeficiency virus (HIV) infection (and other cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary, congenital or acquired immunodeficiencies)
11. Patients with auto-immune disease, with the exception of type I diabetes or treated hypothyroidism
12. Patients with interstitial lung disease
13. Patients with active B or C hepatitis
14. Other malignancy: patients will not be eligible if they have evidence of other active invasive cancer(s) (other than NSCLC) within 5 years prior to screening (except appropriately treated non-melanoma skin cancer or localized cervical cancer, or other local tumors considered cured (e.g.localized and presumed cured prostate cancer)
15. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, and which would, therefore, make the patient inappropriate for entry into this study
16. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment
17. Male patients sexually active with a woman of childbearing potential must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator
18. Breastfeeding women
19. Women with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Costantini, Dr, Study Director — OSE Immunotherapeutics
Locations (78):
- United States (10):
  - East Valley Hematology and Oncology medical Group, Burbank, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - BRCR Medical Center, Inc, Boca Raton, Florida
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Meyer Cancer Center, Weill Cornell Medecine, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Robert W. Franz Cancer Center, Portland, Oregon
  - Gesinger Medical Center, Danville, Pennsylvania
  - Millenium Oncology, Houston, Texas
- Czechia (2):
  - Nemocnice Jihlava, Onkologické oddelení, Jihlava
  - Všeobecná Fakultní nemocnice, Prague
- France (24):
  - Institut Saint Catherine, Avignon
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - CHGU Morvan - Brest, Brest
  - Hôpital Louis Pradel, Bron
  - Centre Hospitalier de Cholet, Cholet
  - Hôpital intercommunal de Créteil, Créteil
  - CHU Grenoble, Grenoble
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier du Mans, Le Mans
  - Hopital Albert Calmette, Lille
  - Paoli-Calmettes Institute, Marseille
  - CHU Montpellier, Montpellier
  - Hôpital Emile Muller, Mulhouse
  - Centre Catherine de Sienne, Nantes
  - Hôpital Saint-Louis, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - Hôpital Larrey - CHU de Toulouse, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours, Tours
  - Centre Hospitalier Troyes, Troyes
  - Institut Gustave Roussy (IGR), Villejuif
- Germany (4):
  - Krankenhaus Mehrheit - Kliniken der Stadt Köln - Lungenklinik, Cologne
  - Klinik für Innere Medizin II Hospital Martha-Maria Halle-Dölau gGmbH, Halle
  - Universitätsklinikum Tübingen Medizinische Klinik II, Tübingen
  - Klinik für Innere Medizin II Universitätsklinikum Ulm, Ulm
- Hungary (6):
  - Magyar Honvedseg Egeszsegugyi Kozpont II szamu telephely, Budapest
  - Országos Korányi TBC és Pulmonológiai Intézet XI Tüdőbelosztály, Budapest
  - Országos Korányi TBC és Pulmonológiai Intézet XIV Tüdőbelosztály, Budapest
  - Semmelweis Egyetem Altalanos Orvostudományi Kar Pulmonologiai Klinika, Budapest
  - Csongrad Megyei Mellkasi Betegsegek Szakkorháza I Tüdőosztály, Deszk
  - Matrai Gyogyintézet, Mátraháza
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Campus Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin (Belinson) Medical Center, Petah Tikva
- Italy (13):
  - IRCCS Oncologico Giovanni Paolo II, Bari
  - Unità Operativa di Oncologia dell'Ospedale Vito Fazzi di Lecce, Piazza Muratore, Lecce
  - Oncologia medica, Legnano
  - Azienda USL 2 Lucca - Dipartimento Oncologico, Lucca
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T), Meldola
  - U.O.C. Pneumologia a indirizzo oncologico, Presidio Ospedaliero Monaldi - Azienda Ospedaliera dei Colli - Via Leonardo Bianchi, Napoli
  - Istituto Oncologico Veneto, IRCCS, Padua
  - Ospedale di Perugia - Oncologia medica, Perugia
  - U.O. Oncologia Ospedale Infermi, Rimini
  - UOC di Oncologia Medica, Policlinico Universitario Campus Biomedico, Roma
  - IRCCS Regina Elena National Cancer Institute, Roma
  - Policlinico Santa Maria alle Scotte, Siena
  - Ospedale Civile Maggiore, Verona
- Poland (4):
  - Klinika Onkologii i Radioterapii , Uniwersyteckie Centrum Kliniczne, Gdansk
  - Przychodnia Lekarska "KOMED", Konin
  - Mazowieckie Centrum Leczenia chorób Płuc i Gruźlicy, Otwock
  - Wojewódzki Szpital Zespolony , Oddział Chemioterapii Nowotworów, Torun
- Spain (9):
  - "Complejo Hospitalario Universitario A Coruna (CHUAC)", A Coruña
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital de Mataro, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario La Paz Servicio de Oncología Médica, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda Servicio de Oncología Médica Consultas externas, 2ª planta, Madrid
  - Hospital de Mataro, Mataró
  - Hospital Universitario Carlos Haya, Málaga
- Milton Keynes Hospital, Milton Keynes, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The supporting information as Study Protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR) may be shared with other researchers if OSE Immunotherapeutics agreed and after signature of a confidential agreement between the parties

REFERENCES:
- [Result] Besse B, Felip E, Garcia Campelo R, Cobo M, Mascaux C, Madroszyk A, Cappuzzo F, Hilgers W, Romano G, Denis F, Viteri S, Debieuvre D, Galetta D, Baldini E, Razaq M, Robinet G, Maio M, Delmonte A, Roch B, Masson P, Schuette W, Zer A, Remon J, Costantini D, Vasseur B, Dziadziuszko R, Giaccone G; ATALANTE-1 study group. Randomized open-label controlled study of cancer vaccine OSE2101 versus chemotherapy in HLA-A2-positive patients with advanced non-small-cell lung cancer with resistance to immunotherapy: ATALANTE-1. Ann Oncol. 2023 Oct;34(10):920-933. doi: 10.1016/j.annonc.2023.07.006. Epub 2023 Sep 11. PMID 37704166
- See also: Link to the manuscript (free access) — http://doi.org/10.1016/j.annonc.2023.07.006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Feb 2016 to Apr 2020, patients with advanced NSCLC were recruited in clinics or hospitals specialized in oncology in Europe, US and Israel to prescreen potential patients for HLA-A2 typing (by central lab). Only HLA-A2 positive patients who fulfilled all eligibility criteria were randomized. A total of 219 patients with ICI resistance were randomized, including 118 patients with ICI secondary resistance (disease progression after ICI >= 12 weeks - primary population for efficacy analysis)
Pre-assignment Details: Only patient with HLA-A2 positive phenotype were eligible
Groups:
- OSE2101: Subcutaneous injection at 5 mg, 1 ml every 3 weeks for 6 cycles, then every 8 weeks until 1 year of treatment and therafter every 12 weeks
- Docetaxel or Pemetrexed: Docetaxel by intravenous infusion over 1 hour at 75 mg/m2 every 3 weeks Pemetrexed by intravenous infusion over 10 minutes at 500 mg/m2 every 3 weeks both with premedication according to international guidelines
Period: Overall Study
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Started (Patients with ICI secondary resistance) | 139 | 80
Completed (primary endpoint is overall survival patient completed has been defined as patient deceased at the end of study) | 116 | 65
Not Completed | 23 | 15
Not completed — patient alive at end of study | 22 | 8
Not completed — Withdrawal by Subject | 1 | 7

BASELINE CHARACTERISTICS:
Population: 219 HLA-A2 positive patients with advanced NSCLC who progressed after sequential or concurrent chemotherapy and Immune Checkpoint Inhibitor (either primary or secondary resistance) were randomized. Safety analysis was done in overall population. Primary efficacy analysis was carried out from stratification factor in subgroup of patients with ICI secondary resistance (who had a disease progression after ICI second line > or equal to 12 weeks)
Groups:
- OSE2101: Subcutaneous injection at 5 mg, 1 ml every 3 weeks for 6 cycles, then every 8 weeks until 1 year of treatment and thereafter every 12 weeks
- Total: Total of all reporting groups
Arm/Group | OSE2101 | Docetaxel or Pemetrexed | Total
Number analyzed (Participants) | 139 | 80 | 219
Age, Categorical [Count of Participants; unit: Participants] — Age at study entry Population: Primary efficacy analysis was carried out in the subgroup of patients with ICI secondary resistance defined as as disease progression after ICI second line > or equal to 12 weeks identified from the stratification factor (previous line of ICI). Safety analysis was done in all patients.
  Participants
    All randomized patients with ICI primary and secondary resistance: <=18 years | 0 | 0 | 0
    All randomized patients with ICI primary and secondary resistance: Between 18 and 65 years | 69 | 45 | 114
    All randomized patients with ICI primary and secondary resistance: >=65 years | 70 | 35 | 105
Age, Continuous [Mean (Full Range); unit: years] — Age at study entry Population: Final analysis was carried out in the subgroup of patients with ICI secondary resistance defined as as disease progression after ICI second line > or equal to 12 weeks identified from the stratification factor (previous line of ICI)
  years
    All randomized patients with ICI primary and secondary resistance | 65.3 [41 to 86] | 63.6 [43 to 81] | 64.7 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Primary efficacy analysis was carried out in the subgroup of patients with ICI secondary resistance defined as as disease progression after ICI second line > or equal to 12 weeks identified from the stratification factor (previous line of ICI)/ Safety analysis was done in all patients
  Participants
    All patients with ICI primary and secondary resistance: Female | 40 | 24 | 64
    All patients with ICI primary and secondary resistance: Male | 99 | 56 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data in 11 patients (n=9 in OSE2101 arm, n=2 in docetaxel or pemetrexed arm)
  Participants
    All patients with ICI primary and secondary resistance: number analyzed (Participants) | 130 | 78 | 208
    All patients with ICI primary and secondary resistance: white | 124 | 76 | 200
    All patients with ICI primary and secondary resistance: Black or African American | 4 | 2 | 6
    All patients with ICI primary and secondary resistance: Asian | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 5 | 7
  Czechia | 0 | 1 | 1
  Poland | 1 | 3 | 2
  Italy | 30 | 18 | 31
  Israel | 8 | 3 | 4
  France | 51 | 31 | 46
  Germany | 2 | 3 | 1
  Spain | 33 | 15 | 26
  Hungary | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS defined as the time from randomisation to death from any cause in patients with ICI secondary resistance
Time Frame: Approx. 24 months
Population: OS analysis in patients with ICI secondary resistance defined as disease progression after ICI second line > or equal to 12 weeks (n=118) OS analysis in the ITT population with ICI resistance (primary and secondary resistance) is described in statistical analysis 2 (n=219)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 80 | 38
Months | 11.1 [8.6 to 13.5] | 7.5 [4.7 to 10.3]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority; p < 0.05, t-test, 2 sided — OS in patients with ICI secondary resistance; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.38 to 0.91] — p=0.017
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; OS in the ITT population with ICI resistance (primary and secondary resistance); Test type: Superiority; p = 0.36, t-test, 2 sided; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.62 to 1.19]

2. Secondary Outcome: Post-Progression Survival
Description: Post-progression survival was defined as the time from the earliest date of progression according to RECIST 1.1 until death in patients with ICI secondary resistance
Time Frame: approximately 24 months
Population: Patients with ICI secondary resistance defined as disease progression after ICI second line > or equal to 12 weeks (n=118)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 80 | 38
months | 7.7 [5.6 to 9.7] | 4.6 [3.1 to 5.8]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Post-progression survival in patients with ICI secondary resistance; Test type: Superiority; p = 0.004, t-test, 2 sided; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.27 to 0.79]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Post-progression survival in ITT population with ICI resistance (primary and secondary); Test type: Superiority; p = 0.0035, t-test, 2 sided; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.39 to 0.83]

3. Secondary Outcome: Time to Worsening ECOG PS
Description: Time to Worsening ECOG PS was defined as the time from randomization to the earliest date when ECOG PS was >1 in patients with ICI secondary resistance. Time to worsening ECPG PS was summarized by treatment arm using the Kaplan-Meier method. The median event time for each treatment arm and the corresponding 2-sided 95% confidence interval were provided. By protocol, ECOG PS was not collected when a patient permanenetly discontinued the study treatment. Patients without ECOG PS worsening were censored at the last time when an ECOG value was recorded.
Time Frame: Approx. 24 months
Population: Patients with ICI secondary resistance
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 80 | 38
months | 9.0 [6.3 to 9.9] | 3.3 [2.3 to 6.7]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Time to worsening ECOG PS >1 in patients with ICI secondary resistance; Test type: Superiority; p = 0.006, t-test, 2 sided; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.23 to 0.80]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Time to worsening ECOG PS in the ITT population with ICI resistance (primary and secondary); Test type: Superiority; p = 0.02, t-test, 2 sided; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.35 to 0.92]

4. Secondary Outcome: Mean Changes in Functional Subscales of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30) From Baseline to Treatment Discontinuation in Patients With ICI Secondary Resistance
Description: Mean change from baseline to treatment discontinuation in Quality of Life (QoL) score of the following functional subscales analyzed separately: global health status, physical, role, cognitive, emotional and social functioning. Each score range from 0 to 100 after normalisation. Highest scores correspond to a better quality of life. The mean score change was assessed using a mixed-effects model for repeated measures analysis with the patient as the random effect, treatment, visit and treatment-by-visit interaction as explanatory variables and baseline score as covariates. If the mean score change is negative, it means a deterioration of QoL. If the mean score change is positive or 0, it means an improvement or stability of QoL
Time Frame: Approx. 24 months
Population: Patients with ICI secondary resistance
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 70 | 25
score on a scale
  Global Health Status | 0.77 [-2.92 to 4.47] | -6.19 [-11.83 to -0.55]
  Physical functioning | -2.74 [-6.21 to 0.73] | -8.75 [-14.17 to -3.33]
  Role functioning | -5.09 [-10.60 to 0.43] | -16.78 [-25.29 to -8.28]
  Emotional functioning | 0.50 [-3.29 to 4.28] | -2.75 [-8.63 to 3.12]
  Cognitive functioning | -3.20 [-7.18 to 0.78] | -7.64 [-13.86 to -1.43]
  Social funtioning | -3.82 [-8.30 to 0.66] | -10.43 [-17.23 to -3.64]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ C30 Global Health Status in Patients with ICI secondary resistance; Test type: Superiority; p < 0.05, Mixed Models Analysis; P Value = 0.045
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Physical functioning in patients with ICI secondary resistance; Test type: Superiority; p = 0.07, Mixed Models Analysis; P Value = 0.07
Statistical Analysis 3: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Role functioning in patients with ICI secondary resistance; Test type: Superiority; p < 0.05, Mixed Models Analysis; P Value = 0.03
Statistical Analysis 4: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Emotional functioning in patients with ICI secondary resistance; Test type: Superiority; p = 0.36, Mixed Models Analysis; P Value = 0.36
Statistical Analysis 5: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Cognitive functioning in patients with ICI secondary resistance; Test type: Superiority; p = 0.24, Mixed Models Analysis; P Value = 0.24
Statistical Analysis 6: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — QLQ-C30 Social functioning; p = 0.11, Mixed Models Analysis; P Value = 0.11

5. Secondary Outcome: Mean Changes in Symptoms Subscales of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30) From Baseline to Treatment Discontinuation in Patients With ICI Secondary Resistance
Description: Mean change from baseline to treatment discontinuation in Quality of Life (QoL) score of the following symptoms subscales analyzed separately: Fatigue, Constipation, Dyspnea, Nausea and Vomiting, Pain, Insomnia, Appetite loss, Diarrhea, Financial Difficulties. Each score range from 0 to 100 after normalisation. Lowest scores correspond to a better QoL. The mean score change was assessed using a mixed-effects model for repeated measures analysis with the patient as the random effect, treatment, visit and treatment-by-visit interaction as explanatory variables and baseline score as covariates. If the mean score change is negative, it means a deterioration of QoL. If the mean score change is positive or 0, it means an improvement or stability of QoL.
Time Frame: Approx. 24 months
Population: QLQ-C30 Symptoms score changes from baseline in patients with ICI secondary resistance
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 70 | 25
score on a scale
  Fatigue | 4.47 [0.21 to 8.72] | 11.95 [5.44 to 18.46]
  Constipation | -5.57 [-9.50 to -1.64] | 7.84 [1.97 to 13.71]
  Dyspnea | 3.99 [-1.26 to 9.24] | 2.77 [-5.24 to 10.77]
  Nausea and Vomiting | -1.49 [-3.83 to 0.84] | 1.21 [-2.37 to 4.80]
  Pain | 4.23 [-0.73 to 9.19] | 0.71 [-7.01 to 8.43]
  Insomnia | 0.42 [-4.25 to 5.08] | -0.29 [-7.24 to 6.65]
  Appetite loss | 0.08 [-4.79 to 4.94] | -2.33 [-9.66 to 4.99]
  Diarrhea | -4.12 [-7.85 to -0.38] | -3.85 [-9.33 to 2.16]
  Financial difficulties | 2.22 [-2.15 to 6.59] | 5.82 [-0.82 to 12.45]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Fatigue in ICI secondary resistance; Test type: Superiority; p = 0.06, Mixed Models Analysis; P Value = 0.06
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Constipation in ICI secondary resistance; Test type: Superiority; p = 0.0003, Mixed Models Analysis; P Value = 0.0003
Statistical Analysis 3: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Dyspnea in ICI secondary resistance; Test type: Superiority; p = 0.80, Mixed Models Analysis; P Value = 0.80
Statistical Analysis 4: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Nausea and Vomiting in ICI secondary resistance; Test type: Superiority; p = 0.21, Mixed Models Analysis; P Value = 0.21
Statistical Analysis 5: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Pain in ICI secondary resistance; Test type: Superiority; p = 0.45, Mixed Models Analysis; P Value = 0.45
Statistical Analysis 6: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Insomnia in ICI secondary resistance; Test type: Superiority; p = 0.87, Mixed Models Analysis; P Value = 0.87
Statistical Analysis 7: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Appetite loss in ICI secondary resistance; Test type: Superiority; p = 0.59, Mixed Models Analysis; P Value = 0.59
Statistical Analysis 8: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Diarrhea in ICI secondary resistance; Test type: Superiority; p = 0.88, Mixed Models Analysis; P Value = 0.88
Statistical Analysis 9: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-C30 Financial difficulties in ICI secondary resistance; Test type: Superiority; p = 0.37, Mixed Models Analysis; P Value = 0.37

6. Secondary Outcome: Mean Changes in Symptoms Subscales of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Lung Cancer (QLQ-LC13) From Baseline to Treatment Discontinuation in Patients With ICI Secondary Resistance
Description: Mean change from baseline to treatment discontinuation in Quality of Life (QoL) score of the following symptoms subscales analyzed separately: Alopecia, Peripheral Neuropathy, Sore mouth, Dysphagia, Dyspnea, Pain in arm or shoulder, Pain in chest, Pain in other parts, Hemoptysis, Coughing. Each score range from 0 to 100 after normalisation. Lowest scores correspond to a better QoL. The mean score change was assessed using a mixed-effects model for repeated measures analysis with the patient as the random effect, treatment, visit and treatment-by-visit interaction as explanatory variables and baseline score as covariates. If the mean score change is negative, it means a deterioration of QoL. If the mean score change is positive or 0, it means an improvement or stability of QoL.
Time Frame: Approx. 24 months
Population: QLQ-LC 13 symptoms score changes from baseline in patients with ICI secondary resistance
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 70 | 25
units on a scale
  Alopecia | 0.44 [-4.74 to 5.63] | 25.83 [17.52 to 34.14]
  Peripheral neuropathy | 2.65 [-2.33 to 7.63] | 13.23 [5.37 to 21.08]
  Sore mouth | 0.82 [-2.27 to 3.91] | 8.52 [3.69 to 13.35]
  Dysphagia | 0.44 [-2.49 to 3.37] | 7.41 [2.85 to 11.98]
  Dyspnea | 4.99 [0.87 to 9.11] | 5.19 [-1.57 to 11.95]
  Pain in arm or shoulder | 5.00 [0.60 to 9.39] | 1.16 [-5.70 to 8.02]
  Pain in chest | 1.61 [-2.38 to 5.60] | -1.37 [-7.61 to 4.86]
  Pain in other parts | 8.17 [1.98 to 14.37] | 6.56 [-3.04 to 13.17]
  Hemoptysis | 0.05 [-1.61 to 1.71] | -1.84 [-4.44 to 0.75]
  Coughing | -3.62 [-8.85 to 1.61] | -6.67 [-14.92 to 1.58]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Alopecia in ICI secondary resistance; Test type: Superiority; p < 0.0001, Mixed Models Analysis; P Value = 0.0001
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC 13 Peripheral neuropathy in ICI secondary resistance; Test type: Superiority; p = 0.03, Mixed Models Analysis; P Value = 0.03
Statistical Analysis 3: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Sore mouth in ICI secondary resistance; Test type: Superiority; p = 0.01, Mixed Models Analysis; P Value = 0.01
Statistical Analysis 4: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Dysphagia in ICI secondary resistance; Test type: Superiority; p = 0.01, Mixed Models Analysis; P Value = 0.01
Statistical Analysis 5: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Pain in arm and shoulder; Test type: Superiority; p = 0.35, Mixed Models Analysis; P Value = 0.35
Statistical Analysis 6: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Pain in chest in ICI secondary resistance; Test type: Superiority; p = 0.43, Mantel Haenszel; P Value = 0.43
Statistical Analysis 7: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Pain in other parts; Test type: Superiority; p = 0.78, Mixed Models Analysis; P Value = 0.78
Statistical Analysis 8: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC 13 Hemoptysis in ICI secondary resistance; Test type: Superiority; p = 0.23, Mixed Models Analysis; P Value = 0.23
Statistical Analysis 9: Comparison: OSE2101 vs Docetaxel or Pemetrexed; QLQ-LC13 Coughing in ICI secondary resistance; Test type: Superiority; p = 0.54, Mixed Models Analysis; P Value = 0.54

7. Secondary Outcome: Disease Control Rate (DCR) at 6 Months
Description: DCR at 6 months defined as the number of patients with Complete Response (CR), Partial Response (PR) or Stable Disease (SD) assessed by investigator per "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions based on CT scan in patients with ICI secondary resistance. Complete Response (CR) defined as disappearance of all target lesions; Partial Response (PR) as >=30% decrease in the sum of the longest diameter of target lesions; Stable disease (SD) defined as neither sufficient shrinkage (compared to baseline) to qualify for CR or PR nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD) (e.g. decrease of the sum of the longest diameters of target lesions <30% or increase up to 20%)
Time Frame: Approx. 6 months
Population: 116 out of 118 patients had measurable lesions per RECIST 1.1 at baseline (n=78/80 in OSE2101 arm, 38/38 in docetaxel or pemetrexed arm). One patient had no post-baseline RECIST 1.1 assessement (n=1 in OSE2101 arm).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 78 | 38
percentage of participants | 24.7 [15.6 to 35.8] | 23.7 [11.4 to 40.2]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; DCR at 6 months in patients with ICI secondary resistance; Test type: Superiority; p = 0.87, Mantel Haenszel; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.43 to 2.75]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; DCR at 6 months in ITT patients with ICI resistance (primary and secondary); Test type: Superiority; p = 0.37, Mantel Haenszel; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.36 to 1.46]

8. Secondary Outcome: Progression Free Survival (PFS) in Patients With ICI Secondary Resistance
Description: PFS was defined as the time from randomization to the earliest date of progression assessed by investigator per "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions based on CT scan in patients with ICI secondary resistance. Progressive disease (PD) defined as increase of target lesions >=20% taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest)
Time Frame: Approx. 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 80 | 38
Months | 2.69 [1.61 to 2.79] | 2.99 [2.56 to 4.47]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Median PFS in patients with ICI secondary resistance; Test type: Superiority; p = 0.29, t-test, 2 sided; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.82 to 2.0]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Median PFS in ITT patients with ICI resistance (primary and secondary); Test type: Superiority; p < 0.05, t-test, 2 sided; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.18 to 2.28]

9. Other Pre Specified Outcome: Objective Response Rate (ORR) in ICI Secondary Resistance
Description: Objective Response rate (OOR) was defined as number of patients with Complete Response (CR) + Partial Response (PR) assessed by investigator per "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions based on CT scan in patients with ICI secondary resistance. Complete Response (CR) defined as disappearance of all target lesions; Partial Response (PR) as >=30% decrease in the sum of the longest diameter of target lesions. Investigator-assessed ORR was an exploratory endpoint as not relevant as primary, nor secondary endpoints to evaluate a cancer vaccine.
Time Frame: Approx. 24 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 78 | 38
percentage of participants | 7.7 [2.9 to 16.0] | 18.4 [7.7 to 34.3]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — ORR in ICI secondary resistance; p = 0.07, Mantel Haenszel; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.10 to 1.11]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — ORR in ITT population with ICI resistance (primary and secondary); p = 0.002, Mantel Haenszel; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.08 to 0.59]

10. Other Pre Specified Outcome: Percentage of Patients With Objective Response at 6 Months in ICI Secondary Resistance
Description: Duration of Objective Response (OOR) was defined as number of patients with Complete Response (CR) or Partial Response (PR) at 6 months assessed by investigator per "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions based on CT scan in patients with ICI secondary resistance. Complete Response (CR) defined as disappearance of all target lesions; Partial Response (PR) as >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Approx. 6 months
Population: 22 out of 118 patients had an ORR and was analyzed for duration of response (n=7/80 in OSE2101 arm, 15/38 in docetaxel or pemetrexed arm).
Measure: Number (95% Confidence Interval); unit: percentage of with objective response
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 7 | 15
percentage of with objective response | 33.3 [4.6 to 67.6] | 26.8 [1.3 to 67.0]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — Duration of response at 6 months in ICI secondary resistance; p = 0.88, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.25 to 5.30]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — Duration of Response at 6 months in ITT population with ICI resistance (primary and secondary); p = 0.57, Regression, Cox; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.43 to 4.60]

11. Other Pre Specified Outcome: Time to Next Lung Cancer Therapy in ICI Secondary Resistance
Description: Time to next lung cancer therapy was defined as the time from randomisation to the date of initiation of the first lung cancer therapy during the survival follow-up form
Time Frame: Approx. 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
Number analyzed (Participants) | 80 | 38
months | 5.4 [4.8 to 7.7] | 9.4 [6.3 to 14.1]
Statistical Analysis 1: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — Time to next lung cancer therapy in ICI secondary resistance; p = 0.04, Regression, Cox; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [1.03 to 3.31]
Statistical Analysis 2: Comparison: OSE2101 vs Docetaxel or Pemetrexed; Test type: Superiority — Time to next lung cancer therapy in ITT population with ICI resistance (primary and secondary); p = 0.02, Regression, Cox; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [1.07 to 2.36]

12. Post Hoc Outcome: Overall Survival Before and During the COVID-19 Period
Description: Survival was assessed from date of randomisation to death in the pre COVID-19 pandemic (patients randomised before february 2019 and followed up to 12 months) and during COVID-19 pandemic (patients randomised after february 2019 and followed up to january 2021)
Time Frame: Approx. 24 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Patients in Pre-COVID-19 Period: All patients randomized before february 2019 and followed up to 12 months
- Patients in the COVID-19 Period: All patients randomised after february 2019 and followed up to january 2021
Arm/Group | Patients in Pre-COVID-19 Period | Patients in the COVID-19 Period
Number analyzed (Participants) | 103 | 116
months | 9.4 [8.0 to 12.2] | 8.1 [6.5 to 9.1]
Statistical Analysis 1: Comparison: Patients in Pre-COVID-19 Period vs Patients in the COVID-19 Period; Test type: Superiority; p < 0.05, t-test, 2 sided; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [1.00 to 1.86]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected in each patient from the date of informed consent' signature until 4 weeks after the last dose of study treatment, up to 24 months
Description: A total of 7 patients did not receive the study treatment (n=1 in OSE2101 arm, n=6 in docetaxel or pemetrexed arm).
Arm/Group | OSE2101 | Docetaxel or Pemetrexed
All-Cause Mortality (participants affected / at risk) | 116/139 | 65/80
Serious Adverse Events (participants affected / at risk) | 47/139 | 33/80
Other Adverse Events (participants affected / at risk) | 125/139 | 67/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSE2101 (N=139) | Docetaxel or Pemetrexed (N=80)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
General physical health deterioration (General disorders) | 4 | 5
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 6 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Giant cell arteritis (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 pneumoniae (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal stenosis (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Balance disorder (Nervous system disorders) | 1 | 0
Brain oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Renal haematoma (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 (0)
Anemiae (Blood and lymphatic system disorders) | 0 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
acute myocardial infarction (Cardiac disorders) | 1 | 0
dysphagia (Gastrointestinal disorders) | 0 | 1
enterocolitis (Gastrointestinal disorders) | 0 | 1
pancreatitis acute (Gastrointestinal disorders) | 1 | 0
gait disturbance (General disorders) | 0 | 1
non cardiac chest pain (General disorders) | 1 | 0
erysipela (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
femur fracture (Injury, poisoning and procedural complications) | 1 | 0
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
aphasia (Nervous system disorders) | 1 | 0
urinary tract obstruction (Renal and urinary disorders) | 0 | 1
acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OSE2101 (N=139) | Docetaxel or Pemetrexed (N=80)
Anemia (Blood and lymphatic system disorders) | 9 | 13
Neutropenia (Blood and lymphatic system disorders) | 0 | 13
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 20 | 14
Diarrhea (Gastrointestinal disorders) | 12 | 21
Vomiting (Gastrointestinal disorders) | 14 | 10
Constipation (Gastrointestinal disorders) | 9 | 11
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 32 | 32
Pyrexia (General disorders) | 24 | 9
Fatique (General disorders) | 13 | 12
Injection site induration (General disorders) | 16 | 0
Chest pain (General disorders) | 13 | 2
Injection site reaction (General disorders) | 13 | 0
Oedema peripheral (General disorders) | 7 | 7
Chills (General disorders) | 9 | 0
Pain (General disorders) | 7 | 5
Injection site pain (General disorders) | 10 | 0
Oedema (General disorders) | 2 | 4
Conjunctivitis (Infections and infestations) | 1 | 5
Weight decreased (Investigations) | 6 | 8
Decreased appetite (Metabolism and nutrition disorders) | 28 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokaliaemia (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Headache (Nervous system disorders) | 7 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 21
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 4
Hypotension (Vascular disorders) | 3 | 4
lacrimation increased (Eye disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
In April 2020 at time of planned interim analysis, decision was taken to prematurely stop the accrual due to COVID-19. Early termination led to small numbers of subject analyzed. The statistical plan was revised to propose the primary efficacy analysis in subgroup of patients with ICI secondary resistance (defined as progression after ICI second line >= to 12 weeks from stratification criteria based on biological and clinical rationale).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT02654587/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02654587/SAP_001.pdf